CLINICAL TRIAL: NCT02001922
Title: COPD Integrated Care Program Valais - Living Well With COPD, a Pilot Study Assessing Feasibility, Acceptability and Effectiveness in the Canton of Valais, Switzerland
Brief Title: Soins intégrés BPCO (Broncho-pneumopathie Chronique Obstructive) en Valais - Mieux Vivre Avec ma BPCO (COPD Integrated Care Program Valais - Living Well With COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier du Centre du Valais (Other)
Collaborators: University of Lausanne Hospitals (Other); Promotion santé Valais (Unknown); Ligue pulmonaire valaisanne (Unknown); Association des médecins de famille du Valais (Unknown); Fondation Bangarter (Other); Swiss National Science Foundation (Other); Swiss School of Public Health (personal grant to Isabelle Peytremann-Bridevaux) (Unknown)
Responsible Party: Principal Investigator, Pierre-Olivier Bridevaux, Professor, Centre Hospitalier du Centre du Valais
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: COPD Integrated Care Valais
Record Dates: First submitted 2013-11-08; First posted 2013-12-05 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Pulmonary disease, chronic obstructive; Integrated care; Outcome and process assessment; Quality indicators, Health care; Self-management,; Patient empowerment; Quantitative and qualitative methods
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD integrated care (Experimental): The intervention will target COPD integrated care, and include a combination of patient-related, professional and organizational elements. It will be centered on patients' needs and focus on self-management education, proactive follow-up (scheduled visits and/or phone contacts), team work, healthcare professionals' training, promotion of pulmonary rehabilitation, physical activity and smoking cessation.
  Interventions: Other: COPD integrated care
- Usual care (No Intervention): Usual COPD care

INTERVENTIONS:
Other: COPD integrated care — The intervention will target COPD integrated care, and include a combination of patient-related, professional and organizational elements. It will be centered on patients' needs and focus on self-management education, proactive follow-up (scheduled visits and/or phone contacts), team work, healthcare professionals' training, promotion of pulmonary rehabilitation, physical activity and smoking cessation.
  Arms: COPD integrated care

SUMMARY:
Background: Chronic obstructive pulmonary disease (COPD) is a progressive respiratory disorder characterized by acute exacerbations that contribute to physical impairment and increased healthcare use and costs. Given the increasing burden of this disease in terms of morbidity, disability, mortality and costs, innovative care models centered on patients and aiming at improving quality and comprehensiveness of care are needed. Effective implementation and evaluation of chronic disease management - integrated care(CDM-IC) programs, in the real world context is of great importance.

Aim of the pilot study: To conduct a pilot study assessing the acceptability, feasibility and effectiveness of a community-based CDM-IC program for COPD patients residing in the canton of Valais.

Design: The evaluation plan of this study will combine both quantitative (controlled before-after study design) and qualitative methods (focus groups with COPD patients and practicing healthcare professionals).

Setting: French-speaking part of the canton of Valais.

Patients: 50 adult (>35 years) COPD patients GOLD stage I (symptomatic) - IV of the disease, non-institutionalized and residing in the canton of Valais. The control group of patients will be constituted of age and gender-matched COPD patients from the Swiss COPD cohort study.

Measures:

Quantitative part:

Primary outcomes: Generic and disease-specific health-related quality-of-life and all-cause hospitalizations (past 12 months)

Other outcomes:

1. Processes of care
2. Patients' assessment of how care is congruent with the Chronic Care Model (PACIC instrument)
3. Measure of self-efficacy (intermediary outcome)
4. 6-minutes walking test, nb of COPD exacerbations, % of current smokers
5. Healthcare utilization: unscheduled ambulatory care visits
6. Care satisfaction
7. Measures of the process of implementation of the intervention

Qualitative part: At 12 months: conduct of two focus groups of participating COPD patients, and of two focus groups of participating healthcare professionals.

DETAILED DESCRIPTION:
Background: Chronic obstructive pulmonary disease (COPD) is a progressive respiratory disorder characterized by acute exacerbations that contribute to physical impairment and increased healthcare use and costs. Given the increasing burden of this disease in terms of morbidity, disability, mortality and costs, innovative care models centered on patients and aiming at improving quality and comprehensiveness of care are needed. Effective implementation and evaluation of chronic disease management - integrated care(CDM-IC) programs, in the real world context is of great importance.

Aim of the pilot study: To conduct a pilot study assessing the acceptability, feasibility and effectiveness of a community-based CDM-IC program for COPD patients residing in the canton of Valais.

Design: The evaluation plan of this study will combine both quantitative and qualitative methods. A controlled before-after study design will be considered for the quantitative part of the project, and the qualitative part will include the conduct of focus groups with COPD patients and practicing healthcare professionals.

Setting: French-speaking part of the canton of Valais.

Patients: 50 adult (>35 years) COPD patients GOLD stage I (symptomatic) - IV of the disease, aged > 35 years, non-institutionalized and residing in the canton of Valais. Patients will be recruited by primary care and pulmonary care physicians practicing in the French-speaking part of the canton of Valais. The control group of patients will be constituted of age and gender-matched COPD patients already included in the Swiss COPD cohort study.

Measures:

Quantitative part:

Primary outcomes: Generic and disease-specific health-related quality-of-life(Chronic Respiratory Questionnaire (CRQ), SF-36 and COPD Assessment Test (CAT)) and all-cause hospitalizations (past 12 months)

Other outcomes:

1. Processes of care (% patients having participated to self-management education sessions, % patients having received/used the action plan, % patients having received smoking cessation recommendations, % patients having received advices/participated to participate to pulmonary rehabilitation, % patients having received influenza immunization during the past 12 months, % patients receiving appropriate treatment, nb of consultations with primary care physician/pulmonary care physician/other, nb of contacts with the hotline)
2. Patients' assessment of how care is congruent with the Chronic Care Model (PACIC instrument)
3. Measure of self-efficacy (intermediary outcome)
4. Health behaviors, symptoms and physical activity measures: 6-minutes walking test, nb of COPD exacerbations during past (past 12 months), % of current smokers
5. Healthcare utilization: unscheduled ambulatory care visits
6. Care satisfaction
7. Measures of the process of implementation of the intervention (nb of recruiting practices and physicians, nb of participating practices and physicians, nb of and patients, of drop-outs, satisfaction of healthcare professionals towards COPD program)

Qualitative part: conduct of two focus groups of participating COPD patients, and of two focus groups of participating healthcare professionals, 12 months after the start of the recruitment.

Development and implementation of the intervention:

The development of the current COPD program in Valais is being implemented in collaboration with physicians working in private practices (family physicians and specialists), physiotherapists, pharmacists and nurse specialists. It will involve academic and public institutions, as well as practitioners. The program has been launched in March 2013, after a preliminary phase involving the conduct of focus groups. Their aims were to explore the needs and barriers to better care, as well as the shape of the targeted CDM elements for better implementation in real life, from the point of view of COPD patients and healthcare professionals.

The CDM intervention considered in the "Soins intégrés BPCO en Valais - Mieux vivre avec ma BPCO" program is based on the " Living well with COPD programme " developed by Prof. Bourbeau & al at McGill University, Montreal, Canada. The "Soins intégrés BPCO en Valais - Mieux vivre avec ma BPCO" program will include a combination of patient-related, professional and organizational elements. It will be centered on patients' needs and focus on self-management education, proactive follow-up (scheduled visits and/or phone contacts), team work, healthcare professionals' training, and promotion of pulmonary rehabilitation, physical activity as well as smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (GOLD stage 1-symptomatic to 4)
* Age >= 35 years
* Residing in the canton of Valais Switzerland, non-institutionalized
* Informed consent

Exclusion Criteria:

* Hospitalization during previous 4 weeks
* Pulmonary rehabilitation during past 18 months
* Estimated life expectancy < 12 months
* Obvious cognitive impairment
* Not speaking or understanding French well enough

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Generic and disease-specific health-related quality-of-life (Chronic Respiratory Questionnaire (CRQ), SF-36, COPD Assessment Test (CAT)) | 12 months
All-cause hospitalizations (past 12 months) | 12 months

SECONDARY OUTCOMES:
Processes of care, patient assessment of chronic illness care (PACIC) | 12 months
6-minutes walking test | 12 months
COPD exacerbations | 12 months
% smokers | 12 months

OTHER OUTCOMES:
Self-efficacy | 12 months
Healthcare utilization | 12 months
Care satisfaction | 12 months
Process of implementation of the intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Peytremann-Bridevaux, MD, MPH, DSc, Principal Investigator — University of Lausanne Hospitals; Bernard Burnand, MD, MPH, Principal Investigator — University of Lausanne Hospitals; Jean-Marie Tschopp, MD, Principal Investigator — Centre Hospitalier du Centre du Valais; Pierre-Olivier Bridevaux, MD, MSc, Principal Investigator — Centre Hospitalier du Centre du Valais
Locations (1):
- Centre Valaisan de Pneumologie, Centre Hospitalier du Centre du Valais, Crans-Montana, Valais, Switzerland